CLINICAL TRIAL: NCT00340535
Title: Levels of Selected Potentially Carcinogenic Drinking Water Disinfection Byproducts in Whole Blood After Showering
Brief Title: Effect of Genetic Differences on Levels of Water Disinfection Byproducts in Blood After Showering
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904228; 04-C-N228; NCT00559793 (obsolete NCT alias); NCT01338272 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Normal Physiology
Keywords: Disinfection byproducts; Genetic Variation; Trihalomethanes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Individuals: Individuals recruited at U of Pittsburgh

SUMMARY:
This study will examine whether genetic differences among individuals affect blood levels of certain chemicals called DBPs after showering. Chemicals such as chlorine and ozone are used to kill germs in water. These chemicals may react with organic matter in the water and form other chemicals called disinfection byproducts, or DBPs. Although people are usually exposed to DBPs by drinking tap water, these chemicals may also penetrate the body during showering. This study will see whether the levels of DBPs after showering vary among individuals depending on differences in genes that code for enzymes called GSTT1, CYP2D6, and CYP2E1, which break down DBPs. This study, sponsored by the Centers for Disease Control and Prevention and the National Institutes of Health, is conducted at the University of Pittsburgh's Center for Clinical Pharmacology.

Healthy adults between 18 and 45 years of age who do not smoke cigarettes and are not taking any medicines may be eligible for this study. Candidates are screened with a medical history and blood and urine tests. Participants are given a diary to record the foods they eat and how much water they drink during the 2 days before their study appointment. The following activities are scheduled on the appointment day:

* Measurements of blood pressure, height, and weight, and pregnancy test for women
* Questions about alcohol consumed and medications taken in the last 48 hours
* Review of food and water diary
* Interview for demographic information (name, address, date of birth, etc.) and other information, such as sex, height, weight. Subjects are also asked about anything, such as exercise, that might affect their breathing, since breathing problems are a rare side effect of chlorzoxazone, a drug used in this study.
* Urine sample collection
* Blood draw and insertion of a small catheter (plastic tube) to allow for additional blood draws during the test procedure without having repeated needle sticks
* 10-minute shower in a private bathroom
* Blood sample collection 10 minutes after the shower and again at 30 minutes after the shower
* Dose of chlorzoxazone (a drug used to treat muscle pain)
* Interview about subject's exposure to water
* Light breakfast
* Blood and urine collections 2 hours after the chlorzoxazone dose
* Lunch
* Observation for drug side effects for 2 hours, or longer if needed

Seven blood samples totaling 75 milliliters (about 5 tablespoonfuls) of blood are collected during this study. The blood is tested for chemicals called trihalomethanes to see how they are broken down. The urine samples are tested for chemicals called haloacetic acids, which are found in tap water after it has been treated with chlorine.

DETAILED DESCRIPTION:
Disinfection byproducts in drinking water (DBP) are inadvertently created when chlorine interacts with organic compounds in the untreated water. DBP have been implicated in elevated risk of several types of cancer. Until recently, ingestion was considered to be the major route of exposure. However, an NCI collaborative study in Spain is now showing a link between bladder cancer and exposure to DBP in water during showering or bathing. However, little is known of the mechanisms of action. Almost all drinking water disinfected with chlorine contains measurable levels of DBP. The DBP found in greatest concentration are the trihalomethanes [(THM); chloroform, bromoform, bromodichloromethane, and dibromochloromethane]. Previously, our collaborators from the CDC measured changes in blood THM levels after showering and bathing, and ingesting water. Showering resulted in the largest increases, with a wide range in the increase among subjects with similar exposures. Enzyme variants due to genetic polymorphisms may be responsible for these differences.

We plan to assess the association between the presence of enzyme variants (genetic polymorphisms) and the increase of trihalomethanes in the blood of people exposed to DBP while showering. The study will be conducted at the General Clinical Research Center (GCRC), Center for Clinical Pharmacology (CCP), University of Pittsburgh, Dr. Robert Branch, Director. Approximately 250 volunteers will be identified from Dr. Branch's ongoing research program. These subjects will have been pre-screened with a normal standard blood panel and for genetic polymorphisms of interest. From this pool of pre-screened individuals, we will recruit approximately 100 people who have enzyme variants of differing activity.

We will ask the 100 volunteers to provide seven 10-mL blood samples and two urine samples, and take a 10-minute shower at the study site (the CCP in Pittsburgh, PA). Blood samples will be analyzed for trihalomethane concentrations, and red blood cell enzyme activities. To study the activity of the enzyme CYP2E1, we will administer a single dose of chlorzoxazone, a muscle relaxant metabolized by this enzyme. We will measure enzyme activity by analyzing blood samples collected 2 hours post-administration. We will conduct a brief interview with each volunteer to obtain demographic and other information that might impact the dose of THM. We will collect ambient air samples before, during and after showering for each participant and analyze them for levels of THMs. A water sample will be collected during showering and analyzed for levels of THM and haloacetic acids. We will ask 10 randomly selected study subjects to repeat study activities for quality control purposes.

Levels of THM in blood before and after showering, and the rate of decrease in blood concentration, will be analyzed with respect to the presence of genetic polymorphisms for selected enzymes, or their phenotypic activity. Blood THM levels will also be compared with various demographic and physiologic measurements. To test intra-individual variation in several measures, ten randomly selected participants (stratified by sex, i.e. 5 males and 5 females) will be asked to conduct the study twice, with the two study appointments separated by at least a week.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will be comprised of non-smoking males and females in the age range 18-45 years. The age range was selected to limit variability in activity of important enzyme systems.

EXCLUSIONS CRITERIA:

Persons with lung conditions will be excluded because inhalation is a major route of exposure for trihalomethanes.

Liver conditions will be excluded because of the potential risks possibly associated with chlorzoxazone administration.

Pregnant and lactating women will be excluded from participation in the study, for multiple reasons, the major one being possible (but unknown) adverse health risks from chlorzoxazone exposure.

In addition, we will exclude persons with chronic conditions such as diabetes who chronically use medication, such as Orinase or others. These persons will be excluded due to unknown effects of such disease on the enzyme systems under investigation and to avoid any possible adverse effects of the study, including chlorzoxazone administration.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: convenience sample of individuals recruited at the University of Pittsburgh.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-06-23 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Blood trihalomethane levels | Before and after showering
  Levels of triahlomethane levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beane-Freeman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Boorman GA. Drinking water disinfection byproducts: review and approach to toxicity evaluation. Environ Health Perspect. 1999 Feb;107 Suppl 1(Suppl 1):207-17. doi: 10.1289/ehp.99107s1207. PMID 10229719
- [Background] Cantor KP, Hoover R, Hartge P, Mason TJ, Silverman DT, Altman R, Austin DF, Child MA, Key CR, Marrett LD, et al. Bladder cancer, drinking water source, and tap water consumption: a case-control study. J Natl Cancer Inst. 1987 Dec;79(6):1269-79. PMID 3480378
- [Background] McGeehin MA, Reif JS, Becher JC, Mangione EJ. Case-control study of bladder cancer and water disinfection methods in Colorado. Am J Epidemiol. 1993 Oct 1;138(7):492-501. doi: 10.1093/oxfordjournals.aje.a116883. PMID 8213753